CLINICAL TRIAL: NCT06205381
Title: A Phase 1, Single And Multiple Ascending Dose, Food Effect, and Drug-Drug Interaction Study With Itraconazole, Midazolam and Fexofenadine Of Orally Administered AV078 In Healthy Adults
Brief Title: Assessment of the Safety, Tolerability and Pharmacokinetics of AV078 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aeovian Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-078-101
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: Healthy Participants
Keywords: mTOR
MeSH Terms: interventions — Itraconazole; Midazolam; fexofenadine

STUDY DESIGN:
Intervention Model Description: Part A will study single doses of AV078 in a double-blind randomized, placebo-controlled, parallel-group and dose-escalating design ("single ascending dose [SAD] study").
  Part B will study repeated doses of AV078 (once daily for 14 days) in a double-blind, randomized, placebo-controlled, parallel-group and dose-escalating design ("multiple ascending dose [MAD] study").
  Part C will study the effect of food on the PK of AV078 in an open-label, randomized sequence 2-way crossover design.
  Part D will study the effect of itraconazole on the PK of AV078 in an open-label, fixed sequence design.
  Part E will study the effect of AV078 on the PK of midazolam and fexofenadine in an open-label, fixed sequence design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Parts A and B of the study comparing AV078 to placebo will be a double-blind design (participant and investigator) Parts C, D and E are open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- AV078 (Experimental): In part A, a single ascending doses of AV078 oral solution will be investigated in separate cohorts. The starting dose will be 0.5 mg and ascending doses will be determined based on data from previous cohorts.
  In Part B, multiple ascending doses of AV078 oral solution will be administered once daily for 14 days. Dose levels will be determined based on data from the single ascending dose study and previous cohorts in the multiple ascending dose study.
  In Part C the effect of food (fasting or high calorie) on the pharmacokinetics of a single dose of AV078 will be investigated. The dose will be determined from Part A of the study.
  Interventions: Drug: AV078
- Placebo (Placebo Comparator): In Part A, placebo oral solution (containing no active ingredient) will be administered once.
  In Part B, placebo oral solution (containing no active ingredient) will be administered once daily for 14 days.
  Interventions: Drug: Placebo
- Itraconazole (Other): In Part D, 200 mg itraconazole will be administered as an oral capsule once daily for 9 days, to investigate the effect of itraconazole on the pharmacokinetics of AV078.
  Interventions: Drug: Itraconazole
- Midazolam and fexofenadine (Other): In Part E, 2.5 mg midazolam will be administered as an oromucosal solution and 120 mg fexofenadine will be administered as an oral tablet on day 1 and day 18, to investigate the effect of AV078 on the pharmacokinetics of midazolam and fexofenadine.
  Interventions: Drug: Midazolam; Drug: Fexofenadine

INTERVENTIONS:
Drug: AV078 — Oral solution containing active ingredient, AV078
  Arms: AV078
Drug: Placebo — Oral solution with no active ingredients
  Arms: Placebo
Drug: Itraconazole — Once daily oral dose of 200 mg itraconazole administered for 9 days
  Arms: Itraconazole
Drug: Midazolam — 2.5 mg midazolam administered orally on day 1 and day 18
  Arms: Midazolam and fexofenadine
Drug: Fexofenadine — 120 mg fexofenadine administered orally on day 1 and day 18
  Arms: Midazolam and fexofenadine

SUMMARY:
This Phase 1 study in healthy adult volunteers is planned to evaluate the safety, tolerability, and pharmacokinetics (PK) of AV078, a selective inhibitor of mammalian target of rapamycin complex 1 (mTORC1).

The study will begin with a standard exploration of safety and tolerability in sequential single ascending dose (SAD) and multiple ascending dose (MAD) cohorts. Subsequent cohorts will collect PK data to evaluate food effects and potential drug-drug interactions relevant to AV078.

DETAILED DESCRIPTION:
This Phase 1 study in healthy adult volunteers is planned to evaluate the safety, tolerability, and pharmacokinetics (PK) of AV078, a selective inhibitor of mammalian target of rapamycin complex 1 (mTORC1). The study will additionally explore the relationship between AV078 and pharmacodynamic biomarkers related to mTOR.

The study will begin with a standard exploration of safety and tolerability in sequential single ascending dose (SAD) and multiple ascending dose (MAD) cohorts, incorporating reviews by a dedicated Safety Review Group to guide dose escalation decisions. The study will also include a cohort using a 2-way crossover design to evaluate food effects on the PK of AV078. The study will additionally include cohorts evaluating potential drug-drug-interactions (DDIs) using coadministration of index substrates and index perpetrators typically used in DDI studies of the relevant enzymes. Specifically, one DDI cohort will assess the effects of administration of itraconazole (a strong inhibitor of CYP3A4) on the PK of AV078, and an additional DDI cohort will assess the effects of administration of AV078 on the PK of midazolam (a sensitive probe substrate for CYP3A4) and fexofenadine (a probe substrate for P-gp).

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy male or female as determined by medical evaluation including medical history, psychiatric history, and no clinically significant findings on physical examination, laboratory tests, and cardiac monitoring. Slight excursions outside of normal limits may be allowed provided they are considered not clinically significant by the investigator.
2. Ages 18-65 years (inclusive), at the time of consent.
3. At least 45 kg with a body mass index (BMI; Quetelet index) in the range 18.0-32.0, at screening.
4. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
5. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or their delegate.
6. Agree not to donate blood or blood products during the study and for up to 3 months after the last administration of the trial medication.
7. Have received at least 2 doses of the COVID vaccine (1 dose of the Janssen-Cilag vaccine is acceptable).

Key Exclusion Criteria:

1. Current, or past history of any clinically significant mental or physical illness or condition that the Investigator concludes would create significant concern for participation in the study.
2. Surgery (eg stomach bypass) or medical condition that might affect absorption of medicines (cholecystectomy is allowed).
3. Presence or history of severe adverse reaction to any drug or a history of sensitivity to midazolam (Part E only), fexofenadine (Part E only) and itraconazole (Part D only), or any excipients in the tablets/solutions.
4. History of relevant atopy including any confirmed significant allergic reactions against any drug, or multiple drug allergies (non-active hay fever is acceptable)
5. History of suicidal behaviour or express or have any suicidal ideation on the C-SSRS at screening or admission.
6. Employee of the Sponsor, the CRO and/or study site or their relatives.
7. Unable or unwilling to eat a high-fat breakfast per study requirements (Part C only).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs). | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Occurrence of clinically significant changes in physical examination (including neurological assessment). | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Abnormal physical examination findings will be listed.
Change in blood haematology values. | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Haematology data will be summarised by treatment
Change in blood biochemisty values. | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Biochemistry data will be summarised by treatment
Change in urinalysis values. | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Urinalysis data will be summarised by treatment
Change in lipid panel values. | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Lipid panel data will be summarised by treatment
Change in blood coagulation values. | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Blood coagulation data will be summarised by treatment
Clinically significant ECG findings. | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  Occurrence of clinically significant ECG findings will be listed.
Monitor for the emergence of suicidal ideation and behaviour using the Columbia-Suicide Severity Rating Scale (C-SSRS). | From screening (Day -42) to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
  C-SSRS will be listed and summarised for each visit.
Pharmacokinetics measured by area under the concentration-time curve in fasted and fed state. | Day 1 to Day 7 post-dose and final follow-up visit (Day 14)
  To determine the effect of food on the pharmacokinetic profile of AV078.
Pharmacokinetics measured by the maximum plasma concentration (Cmax) in fasted and fed state. | Day 1 to Day 7 post-dose and final follow-up visit (Day 14)
  To determine the effect of food on the pharmacokinetic profile of AV078.
Effects of itraconazole on the pharmacokinetics of AV078 measured by area under the concentration-time curve. | Day 1 to Day 15 post-dose and final follow-up visit (Day 23)
Effects of itraconazole on the pharmacokinetics of AV078 measured by the maximum plasma concentration (Cmax). | Day 1 to Day 15 post-dose and final follow-up visit (Day 23)
Effects of AV078 on the pharmacokinetics of midazolam and fexofenadine measured by area under the concentration-time curve. | Day 1, 2, 18 and 19 post-dose (midazolam) or Day 1-3, 18 and 19 post-dose (fexofenadine)
Effects of AV078 on the pharmacokinetics of midazolam and fexofenadine measured by the maximum plasma concentration (Cmax). | Day 1, 2, 18 and 19 post-dose (midazolam) or Day 1-3, 18 and 19 post-dose (fexofenadine)

SECONDARY OUTCOMES:
Pharmacokinetics of AV078 measured by the area under the concentration-time curve. | Day 1 to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Pharmacokinetics of AV078 measured by the maximum plasma concentration (Cmax). | Day 1 to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Pharmacokinetics of AV078 measured by time of maximum plasma/whole blood concentration. | Day 1 to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Pharmacokinetics of AV078 measured by terminal elimination half-life. | Day 1 to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Pharmacokinetics of AV078 measured by fraction of drug excreted in urine. | Day 1 to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Pharmacokinetics of AV078 measured by renal clearance from plasma/whole blood. | Day 1 to final visit post-treatment (Day 14 for Part A and Day 42 for Part B).
Change from baseline and placebo-corrected change from baseline in ECG parameter, QTcF including exposure response. | Part A: Screening (Day -42) to Day 5 post-dose, and final follow-up visit (Day 14). Part B: Screening (Day -42) to Day 2 post-dose, then Day 4, 7, 10, 14, 15 and 18 post-dose, and final follow-up visit (Day 42)]
Change from baseline and placebo-corrected change from baseline in ECG parameter - heart rate (HR) | Part A: Screening (Day -42) to Day 5 post-dose, and final follow-up visit (Day 14). Part B: Screening (Day -42) to Day 2 post-dose, then Day 4, 7, 10, 14, 15 and 18 post-dose, and final follow-up visit (Day 42)]
  ECG parameters will be descriptively summarised at each time point.
Change from baseline and placebo-corrected change from baseline in ECG parameter - PR interval | Part A: Screening (Day -42) to Day 5 post-dose, and final follow-up visit (Day 14). Part B: Screening (Day -42) to Day 2 post-dose, then Day 4, 7, 10, 14, 15 and 18 post-dose, and final follow-up visit (Day 42)]
  ECG parameters will be descriptively summarised at each time point.
Change from baseline and placebo-corrected change from baseline in ECG parameter - QRS interval | Part A: Screening (Day -42) to Day 5 post-dose, and final follow-up visit (Day 14). Part B: Screening (Day -42) to Day 2 post-dose, then Day 4, 7, 10, 14, 15 and 18 post-dose, and final follow-up visit (Day 42)]
  ECG parameters will be descriptively summarised at each time point.
Incidence and severity of treatment emergent adverse events (TEAEs) | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Assessed for single doses of AV078 taken fasted or after a high-fat breakfast and repeated oral doses of AV078
Occurrence of clinically significant changes in physical examination (including neurological assessment). | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Abnormal physical examination findings will be listed.
Change in blood haematology values | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Haematology data will be summarised by treatment.
Change in blood biochemistry values | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Biochemistry data will be summarised by treatment.
Change in urinalysis values | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Urinalysis data will be summarised by treatment.
Change in lipid panel values | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Lipid panel data will be summarised by treatment.
Change in blood coagulation values | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  Coagulation data will be summarised by treatment.
Monitor for the emergence of suicidal ideation and behaviour using the Columbia-Suicide Severity Rating Scale (C-SSRS) | From screening (Day -42) to final visit post-treatment (Day 14 for Part C, Day 23 for Part D and Day 26 for Part E)
  C-SSRS will be listed and summarised for each visit

CONTACTS AND LOCATIONS:
Overall Officials: Davis Ryman, Study Director — Chief Medical Officer, Aeovian Pharmaceuticals
Locations (2):
- Australia (2):
  - Q-Pharm, Herston, Queensland
  - Nucleus Network Pty Ltd, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No